CLINICAL TRIAL: NCT06500832
Title: An Analysis of Clinicians' Knowledge and Attitudes Regarding Defensive Dentistry Practices: A Survey-based Research
Brief Title: Defensive Dentistry Practices and Dentists (DDP)
Status: Completed | Type: Observational
Sponsor: Istanbul Aydın University (Other)
Responsible Party: Principal Investigator, Asst. Prof. Dr. Suleyman Emre Meseli, Assoc. Prof. Suleyman Emre MESELI, PhD, DDS, Istanbul Aydın University
Other Study IDs: IAUDENT-02
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Defensive Medicine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All participants
  Interventions: Other: Survey-based Data Collection Tool

INTERVENTIONS:
Other: Survey-based Data Collection Tool — The data collection tool to be presented to the participants is planned as a three-part survey. The first part of this form asked 9 questions about the demographic characteristics of the participants consisted of age, gender, marital status, duration in the profession, specialization in dentistry, type of workplace, and off-the-clock work.
  The second part of the data collection tool consisted of the 'Defensive Dentistry Practice Survey,'(DDPS) DDPS which is the original language of which is Turkish, is a 5-point Likert-type scale. A total of 12 statements about DDPS which measure the opinions, attitudes, or behaviors of the participants in terms of DDP, the following options are used: strongly disagreed, disagreed, neither disagreed nor agreed, agreed and strongly agreed, each expressing groups of 20%.
  The last part of the survey had 3 close-ended questions with yes-no options expressing 50% groups is used.

SUMMARY:
Medical malpractice claims have been on the rise in recent years due to the growing patient rights movement. This term is defined as an injury caused by a healthcare professional's failure to follow standard practice during treatment, a lack of skill, or failure to provide treatment. Defensive dentistry is on the rise as violence and malpractice claims increase. Defensive dental practices (DDP) refer to minimize legal responsibility of the clinician primarily rather than looking out for the patient's benefit. This study aims to evaluate the knowledge, awareness and attitudes of dentists in terms of DDP.

ELIGIBILITY:
Inclusion Criteria:

* Having worked as a dentist for at least one year;
* Speaking Turkish as their native language;
* Being a member of the Turkish Dental Association;
* Participating in the study voluntarily.

Exclusion Criteria:

-To stop volunteering until the study is completed.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All participants are the volunteered dentists registered as a member of Turkish Dental Association
Sampling Method: Non-Probability Sample
Enrollment: 410 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
DDPS Score | 1hour
  Total DDPS score of a participant is determined by assigning points as "completely disagreed" (1 point), "disagreed" (2 points), "neither disagreed nor agreed" (3 points), "agreed" (4 points), "completely agreed" (5 points). The total scores are categorized considering the cut-off values as very poor (23-12), poor (35-24), good (47-36), very good (60-48) to determine the level of participants' attitudes towards DDP.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Aydin University, Istanbul, Kucukcekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Baungaard N, Skovvang PL, Assing Hvidt E, Gerbild H, Kirstine Andersen M, Lykkegaard J. How defensive medicine is defined in European medical literature: a systematic review. BMJ Open. 2022 Jan 20;12(1):e057169. doi: 10.1136/bmjopen-2021-057169. PMID 35058268
- [Background] Raposo VL. Defensive Medicine and the Imposition of a More Demanding Standard of Care. J Leg Med. 2019 Oct-Dec;39(4):401-416. doi: 10.1080/01947648.2019.1677273. PMID 31940251